CLINICAL TRIAL: NCT06128187
Title: The Effect of Dual Task Training With Virtual Reality on Upper Extremity Functions and Cognitive Functions in Stroke Patients
Brief Title: The Effect of Dual Task Training on Upper Extremity Functions in Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Muş Alparslan University (Other)
Responsible Party: Principal Investigator, Ramazan Öztürk, physiotherapist, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023/06-69
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: STROKE REHABİLİTATİON
Keywords: Stroke, Rehabilitation, Virtual Reality, Upper Extremity
MeSH Terms: conditions — Stroke | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Two groups. Study group and control group
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants were enrolled in treatment without being aware of differences in treatment between groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Participants will undergo a conventional upper extremity rehabilitation program for 45 minutes daily, 5 days a week, for 6 weeks. After the conventional rehabilitation program, 30 minutes of virtual reality training for the upper extremity will be applied.
  Interventions: Other: Control Group
- Study Group (Active Comparator): Participants will undergo a conventional upper extremity rehabilitation program for 45 minutes a day, 5 days a week, for 6 weeks. In addition to the conventional rehabilitation program, dual-task training will be provided with a 30-minute virtual reality training program. Cognitive tasks will be given in addition to virtual reality training as dual-task training.
  Interventions: Other: Study Group

INTERVENTIONS:
Other: Control Group — Participants will receive treatment 5 days a week, 45 minutes a day for 6 weeks. After the traditional rehabilitation program, 30 minutes of virtual reality training will be given.
  Arms: Control Group
Other: Study Group — Participants will receive treatment 5 days a week, 45 minutes a day for 6 weeks. After the traditional rehabilitation program, 30 minutes of dual-task training will be given
  Arms: Study Group

SUMMARY:
Purpose: To investigate the effect of upper extremity single and double task training using virtual reality on upper extremity functions, cognitive functions and dual task performance in stroke patients. Our aim is to determine the effectiveness of dual-task upper extremity training compared to single-task training.

DETAILED DESCRIPTION:
Purpose: To investigate the effect of upper extremity single and double task training using virtual reality on upper extremity functions, cognitive functions and dual task performance in stroke patients.

Materials and Methods: The study was planned on patients who applied to Erenkoy Physical Therapy and Rehabilitation Hospital and were diagnosed with hemiplegia by a specialist neurologist. Participants who met the inclusion criteria in the study will be divided into two groups as Group 1 = study group and group = 2 control groups by computerized randomization method. For the evaluation of upper extremity functions of the participants whose socio-demographic characteristics were recorded; Fugl Mayer Upper Extremity Assessment Scale, Box and Blocks Test (BBT), Stroop Test and Montreal Cognitive Assessment Scale (MOCA) will be used to evaluate cognitive functions. The Barthel index of daily living activities of the patients and the Stroke-Specific Quality of Life Assessment Scale will be used to evaluate the health-related quality of life. Evaluation of double-task performance will be evaluated by the Box and Blocks Test (BBT) and a cognitive task added to the Xbox 360 Kinect game apps. Participants will be evaluated 4 times before the treatment, after the treatment and at the 1st month and 3rd month after the treatment in order to see the sustainability of the effect of the rehabilitation program.

Patients in both groups will receive a conventional upper extremity rehabilitation program (neurophysiological methods, joint range of motion exercises, strengthening exercises, occupational therapy) and 30 minutes of virtual reality training for 6 weeks, 5 days a week, for 45 minutes daily. Participants in the study group will be given double-task training in addition to stroke rehabilitation and virtual reality training. Dual task training will be performed with the addition of cognitive tasks in addition to virtual reality training.

Cognitive Tasks;

1. Attention-oriented, e.g. Counting numbers: Counting numbers backwards three by three from the participant rhythmically,
2. For memory, e.g. describing activities of daily living: Describing an event from the participant in detail,
3. For executive functions, e.g. Verbal communication: It will be planned in the form of giving the participant a letter from the alphabet and asking for words in certain categories such as plants, animals and countries. As progress is made, the difficulty of the missions will increase.

Xbox 360 Kinect game console will be used for virtual reality treatment. In the treatment, a rehabilitation program will be prepared with games that require complex upper extremity movements such as tennis, golf, darts and boxing to improve upper extremity functions.

We think that dual-task training will increase upper extremity functions and cognitive functions. Due to the lack of dual-task training studies with the upper extremity, we think that our study will contribute to upper extremity rehabilitation protocols and dual-task training literature.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with hemiplegia for the first time
* Patients aged ≥18 years
* Medically stable
* According to Brunnstrom stages, the upper extremity is at stage 3 and above
* Must have the ability to understand, hear and speak sufficiently to perform treatment with a game console.
* Montreal Cognitive Assessment (MoCA) score ≥ 21
* Patients who are literate

Exclusion Criteria:

* Presence of high blood pressure, heart disease, vision problems
* Those with risk of shoulder subluxation and fracture
* Hemiplegic side, with joint movement limitation in the upper extremity Having a history of epileptic seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-11-15 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Box and Block test (BTT) | 18 weeks
  Box and Block test (BBT) was used to measure unilateral gross manual dexterity. This test consists of moving, one by one, the maximum number of blocks from one compartment of a box to another of equal size within 60seconds. The patients had number of blocks moved within 60seconds was recorded. The higher number of blocks moved, the higher score you get.

SECONDARY OUTCOMES:
Fugl-Meyer Assessment (FMA-UL) | 18 weeks
  The upper limb score in the Fugl-Meyer Assessment (FMA-UL) was used for primary outcome measure to assess the motor function of both upper extremities in- cluding the shoulder, elbow, forearm, wrist, and hand. The FMA-UL is widely used for comprehensive clinical examination of arm function, and the maximal score of FMA-UL is 66 points
Barthel index | 18 weeks
  The Barthel scale is an ordinal scale used to measure performance in activities of daily living (ADL). Each performance item is rated on this scale with a given number of points assigned to each level or ranking. It uses ten variables describing ADL and mobility. A higher number is associated with a greater likelihood of being able to live at home with a degree of independence following discharge from hospital.
Stroke Specific Quality Of Life scale (SS-QOL) | 18 weeks
  The Stroke Specific Quality Of Life scale (SS-QOL) is a patient-centered outcome measure intended to provide an assessment of health-related quality of life specific to patients with stroke.
Montreal Cognitive Assessment (MoCA) | 18 weeks
  The MoCA test is a simple, in-office tool that can quickly determine if there is any impairment in a person's cognitive function, including their ability to understand, reason, and remember. The MoCA test is based on scores with a maximum score of 30. The MoCA test examines seven domains (aspects) of cognitive function with a total of 11 different exercises and tasks.
stroop test | 18 weeks
  The Stroop test will used to measure cognitive function in the present study. This test simultaneously reflects reaction time (speed aspect) and accuracy. Here, the effect of different performance levels among the subjects was minimized by specifying the reaction time as the number of items performed within a given time. In addition, accuracy will measured using the number of errors made.
Digit Span Test (DST) | 18 weeks
  Digit Span Test (DST) is a widely-used neuropsychological test in the assessment of attention and working memory, which consists two sections, forward and backward span.
oktem SBST | 18 weeks
  Oktem (SBST) Test is a test that analyzes verbal learning and memory capacity. Information is collected about the participant's instant memory and ability to sustain attention.

CONTACTS AND LOCATIONS:
Overall Officials: Ramazan öztürk, Study Director — Marmara University
Locations (2):
- Turkey (Türkiye) (2):
  - Erenkoy physical therapy and rehabilitation hospital, Istanbul
  - Marmara üniversitesi, Istanbul